CLINICAL TRIAL: NCT04048109
Title: The Point of View of Adolescents Who Have Undergone a Suicidal Act: What Do They Expect from Their Relationship with Their Doctor?
Acronym: Attente_ado
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2019/JLC-02
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Suicidal Act

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Evaluate the expectations of adolescents who have performed a suicidal act with regard to their relationship with their doctor

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who have undergone a suicidal act and who were initially treated by the paediatric emergency department of the University Hospital of Nîmes.
* Teenagers with an attending physician.
* Adolescents who do not object to participating in the study
* Parents (holder of parental authority) who do not object to their child participating in the study
* Preliminary agreement to participate in the research project of the child psychiatrist treating the child.

Exclusion Criteria:

* - Patient who has objected to the use of his data.
* Refusal by the child psychiatrist to participate in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents aged 12 to 18 years with suicidal act
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
percentage of adolescents with poor relationship with the doctor | 2019

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No